CLINICAL TRIAL: NCT00358098
Title: For Women With Estrogen Positive Metastatic Breast Cancer Discordance of Pre-treatment FDG-PET and FES-PET in Addition to Presence of Ki-67 and Human Epidermal Growth Factor 2 (HER-2) Overexpression Will Predict for Hormone Refractory Disease When Compared to Standard Response Criteria
Brief Title: Study to Determine the Utility of FES-PET and FDG-PET in the Prediction of Response to Hormone Therapy in Women With Estrogen Positive Metastatic Breast Cancer
Status: Terminated | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: BR-1-0093
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Breast Cancer
Keywords: PET; hormone positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study of hormone positive (estrogen receptor [ER]), metastatic invasive ductal breast cancer looks at functional scanning using positron emission tomography (PET) and patient response to hormone therapy. Functional scans allow investigators to see more than one metastatic location. The investigators will use an estrogen based agent (FES) to see the number of hormone positive metastases and compare that to positive lesions on routine glucose (FDG) based scanning.

FES and FDG-PET results will be compared to give a FDG to FES ratio. The PET ratio will be calculated before hormone therapy and at relapse after treatment. The investigators will biopsy an accessible lesion that is FDG positive and FES negative and perform pathological testing for ER and PR positivity and compare it to the original primary tumor ER/PR. The investigators will test the lesion for tumor proliferation (using Ki-67) and aggressiveness using human epidermal growth factor receptor 2 (HER-2). Results will be compared to the primary tumor Ki-67 and HER-2 to determine concordance.

The investigators will have pre-treatment results for FES and FDG-PET, will calculate the ratio, and will correlate it to the primary metastatic lesion and test for ER/PR, Ki-67, and HER-2, and subsequent response to therapy. The investigators will determine the FES-PET predictive value for determining appropriateness of hormone therapy for metastatic disease. With these results, the investigators plan to undertake future tumor biomarker/PET studies in metastatic breast cancer.

DETAILED DESCRIPTION:
Primary objective: To determine the utility of pre-treatment (16 alpha[18-F]-fluoroestradiol) FES-PET and routine ([18-F]-fluorodeoxy-D-glucose) FDG-PET in the prediction of response to hormone therapy using standard response criteria (RECIST) as gold standard in 100 primary tumor hormone positive (ER+) women with metastatic carcinoma of the breast.

We will measure standardized uptake ratio (SUV) for FDG and FES at baseline and correlate same to FDG/FES SUV ratio at disease relapse. We predict increased FDG/FES ratio at relapse and using the Pearson correlation coefficient will examine the regression equation slope as a measure of the changing ratio.

Twenty - forty patients will have core biopsy of accessible FDG positive and FES negative metastasis. Metastatic lesion immunohistochemistry (IHC) for ER will be compared to pretherapy FES result for concordance. With 80% agreement level for negative FES and negative core biopsy ER IHC 95% confidence limits (DI) are 56-94% for 20 and 64-90% for 40 patients respectively.

Proliferative index and tumor aggressiveness using IHC for Ki-67 and HER-2 respectively will be measured on primary tumor and biopsied metastatic lesion and correlated with metastatic disease response (RECIST).

Secondary objectives regarding HER-2 and Ki-67 IHC and response will be evaluated using Fisher's exact test for 2 X 2 tables for the 100 women and the 20-40 having core biopsy.

From the sensitivity and specificity determinations, calculated observed agreement between pretherapy FDG FES-PET ratio and RECIST will be 86% (95% CI 78-92%).

Assuming 40% response rate for 100 women receiving first, second or third line hormonal therapy and RECIST response as gold standard, we chose 80% sensitivity (95% CI 64-91%) and 90% specificity (95% CI 80-96%) as giving sufficiently robust data to warrant further studies.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic invasive ductal ER positive breast cancer
* All adjuvant treatment must have been completed at least 3 months prior to study entry.

Exclusion Criteria:

* Patients who do not have the primary tumor subtype of invasive ductal adenocarcinoma
* Patients with only loco-regional recurrence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2006-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Tonkin, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada